CLINICAL TRIAL: NCT06847048
Title: Effects of Using Various Heel-warming Methods Such As Warm Towel Warming and a Thermophore Heating Pad Warming Before Heel Prick on Newborns' Pain Level and Duration of Crying
Brief Title: Nonpharmacological Methods in Heel Stick Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diler Yilmaz (Other)
Responsible Party: Sponsor-Investigator, Diler Yilmaz, Professor, Bandırma Onyedi Eylül University
Organization: Bandırma Onyedi Eylül University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BANU-D-YILMAZ-003
Record Dates: First submitted 2025-02-18; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Pain Management; Newborn Pain
MeSH Terms: conditions — Agnosia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Thermophore pad warming group (Experimental): In the literature, (Lehmann, 1990; Shu et al., 2014), it is recommended that the heel should be warmed at a temperature ranging between 40°C and 45°C to increase blood flow before the heel prick test was performed. During the intervention, the newborn was wrapped with its own blanket leaving the extremity to be treated uncovered. Then, the thermophore heating pad filled with 40°C water was used to warm the sole of the foot for approximately 5 minutes just before the intervention. Attention was paid to prevent the thermophore heating pad from touching other parts of the baby's skin.
  Interventions: Procedure: Thermophore pad warming group
- Warm towel warming group (Experimental): In this group, to warm the heel, the heel area where the blood would be taken was wrapped with a previously heated towel before heel prick. A clean cotton towel was used to warm the newborns' heels. Before the intervention, to warm the towel, it was wrapped in a thermophore pad filled with water at a temperature of approximately 40°C-45°C. The foot area and the heel of the newborn where the blood would be taken were wrapped with a warm towel for 3-4 minutes before heel prick was performed.
  Interventions: Procedure: Warm towel warming group
- Control group (Experimental): In the newborns in this group, heel prick intervention was performed in line with the routine interventions of the clinic. The baby was wrapped in a blanket leaving the foot from which the blood sample would be taken unwrapped.
  Interventions: Other: Control group

INTERVENTIONS:
Procedure: Thermophore pad warming group — Thermophore pad waa using heel warming
  Arms: Thermophore pad warming group
Procedure: Warm towel warming group — In this group, to warm the heel, the heel area where the blood would be taken was wrapped with a previously heated towel before heel prick.
  Arms: Warm towel warming group
Other: Control group — in this group, heel prick intervention was performed in line with the routine interventions of the clinic.
  Arms: Control group

SUMMARY:
In the present study, the randomized controlled and experimental design is used because it was aimed to determine the effects of two different warming methods (warming with a thermophore heating pad and warming with a warm towel) performed before heel prick intervention on pain levels and duration of crying in healthy term newborns.

Study hypotheses are; Hypothesis 1. Using the thermophore pad warming method in newborns before heel prick reduces the newborn's pain level.

Hypothesis 2. Using the warm towel warming method in newborns before heel prick reduces the newborn's pain level.

Hypothesis 3. Using the thermophore pad warming method in newborns before heel prick reduces the duration of crying.

Hypothesis 4. Using the warm towel warming method in newborns before heel prick reduces the duration of crying

DETAILED DESCRIPTION:
Heel prick, intervention performed to take blood sample from the heel, which is frequently performed in newborns, is a more painful intervention than are other methods of taking blood samples. In several studies, it has been indicated that the use of various non-pharmacological methods such as sucrose administration, breastfeeding, skin-to-skin care, acupressure, swaddling, positioning, non-nutritive sucking, foot reflexology, vibration, laser acupuncture, warming the baby's heel reduce infants' pain during heel prick.

This study is a prospective, randomized and controlled trial. In this study aim, was aimed at determining the effects of two different heel warming methods (warming with a thermophore heating pad and warming with a warm towel) performed before heel prick on healthy term newborns' pain levels and duration of cryingin newborns will be examined.

The minimum number of newborns to be included in the study was calculated as 150 using the G*Power (3.1. 9.7) program (margin of error: 5%, confidence interval: 0.95, power: 0.80). The 150 newborns in the sample were randomly assigned into the following three groups in equal numbers via an internet-based program (http://www.randomizer.org): control group (n = 50), thermophore-warming group (n = 47) and warm towel-warming group (n = 50).

Data Collection Tools To collect the study data, the "Descriptive Information Form", "Follow-up Form", and "Neonatal Infant Pain Scale" were used.

ELIGIBILITY:
Inclusion Criteria:

* Having been born at 38-42 weeks of gestation,
* having a birth weight of 2500 g and above,
* having a 5-min APGAR score of 7 and above,
* having stable health,
* having been fed within an hour before the intervention, being calm and not crying before the intervention,
* having a postnatal age of 24-72 hours, and
* undergoing heel prick for the first time

Exclusion Criteria:

* Parents with any mental problems
* Infants with any chronic disease and congenital anomalies.

Ages: 1 Day to 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale (NIPS) | Pain levels of the newborns evaluated during the procedures
  Neonatal Infant Pain Scale: NIPS was developed by Lawrence et al. (1993)21 to evaluate behavioral and physiologic pain responses of preterm and term infants. The scale was adapted to Turkish by Akdovan (1999)22. In the present study, NIPS was used to evaluate the interventional (procedural) pain level of newborns. The scale consists of five behavioral (facial expressions, crying, wakefulness, arm and leg movements) and a physiologic (breathing) signs; 0-2 points are given to the crying indicator, 0-1 points are given to other indicators, and the total score is between 0 and 7. High scores indicate that the severity of pain is excessive.

SECONDARY OUTCOMES:
Total criying time | The time of the procedure was measured from the beginning to the end of the heel stick procedure.
  Duration of crying were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University, Bandirna, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available. I did not find It appropriate to share it.